CLINICAL TRIAL: NCT00507325
Title: Blood and Tumor Sample Collection From Patients With Malignant Melanoma for Long Term Storage
Brief Title: Sample Collection From Melanoma Patients
Status: Terminated | Type: Observational
Why Stopped: Per PI
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-0466
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Melanoma
Keywords: Malignant Melanoma; Blood Sample; Tumor Sample; Long-term storage; Sample Collection
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients will provide blood and tumor samples to help researchers learn about melanoma and other cancers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blood Sample + Tumor Sample: Blood samples will be collected. Tumor samples will be collected using a small needle, a punch knife, or a small surgery.
  Interventions: Procedure: Blood Sample; Procedure: Tumor Sample

INTERVENTIONS:
Procedure: Blood Sample — Blood samples will be collected.
Procedure: Tumor Sample — Tumor samples will be collected using a small needle, a punch knife, or a small surgery.

SUMMARY:
The goal of this laboratory research study is to collect blood and tumor samples from patients with malignant melanoma. Researchers want to store these samples in a secure and confidential laboratory at M. D. Anderson. Researchers will use the information that is learned in this study to help find ways to improve treatment for melanoma and other cancers.

DETAILED DESCRIPTION:
Researchers at M. D. Anderson want to learn as much as possible about melanoma and other cancers. One way researchers can learn more about cancer is by studying what is in your blood and in your tumor.

If you agree to take part in this study, the way you participate will depend on if you are being treated for cancer. If you are receiving any form of chemotherapy, you will have about 4 1/2 tablespoons of blood drawn before you start the first day of treatment. You will then have about 3 tablespoons of blood drawn every 6 to 8 weeks for the next 6 months. You will have a total of up to about 5 blood draws for this portion of the study. You will have the above blood draws during routine visits so that no additional visits will be required.

If you are receiving "immunologic or targeted" cancer treatment, you will have blood drawn for testing. Immunologic treatment is a kind of treatment which boosts your immune system to fight your cancer. Targeted cancer treatment is a kind of treatment which disrupts the functions of proteins that are needed for tumor growth. About 4 1/2 tablespoons of blood drawn before you start the first day of treatment. You will then have about 3 tablespoons of blood drawn 1 time during the first 2 weeks (Days 2-14), 1 time during the second 2 weeks (Days 15-28), 1 time during second or third month (Days 29 - 90), and then once every 3 months for up to 5 years. A total of no more than 25 samples will be drawn.

After the 6-month period, if follow-up is scheduled for you at M. D. Anderson, you will have about 3 tablespoons of blood drawn (during the follow-up visits) once every 3 months for the next 5 years. You will have a total of 20 blood draws for this portion of the study. During your follow-up, you will have a routine clinic visit to monitor any tumor recurrences (occurring again). You will continue to have this visit about every 2 to 6 months, depending on the risk of any tumor recurrence.

If you are not receiving any form of cancer treatment, you will have about 4 1/2 tablespoons of blood drawn on the day that you enroll in this study. If you agree (it is your choice) to participate in the follow-up portion of this study, you will have about 3 tablespoons of blood drawn (during the follow-up visits) once every 3 months for the next 5 years. You will have a total of about 21 blood draws for this portion of the study.

If you do not agree to take part in the additional follow-up, your participation in this study will be over.

If you are planning to have surgery to remove your tumor as part of your standard care, some of your tumor samples will be collected at that time and stored in a secure and confidential laboratory at M. D. Anderson. If the tumor samples are too small, the whole tumor sample will be sent to a doctor for a diagnostic evaluation. If this is the case, researchers will not use any of your tumor sample for this study.

If you have tumors like skin lesions or lymph node lesions that are located close to the skin, and you plan to have cancer treatment, a sample of your tumor will be collected before you receive your cancer treatment. It will also be collected up to 2 other times (for this study's research), while you are on treatment. A total number of biopsy will not exceed 6 per year, and will not exceed more than 10 over 5 year period. The biopsies will be performed by using a small needle (with or without an ultrasound imaging machine), a punch knife, or a small surgery. If you have tumors located close to the skin but do not plan to receive cancer treatment, you will be asked to have a tumor biopsy up to 2 times per year for up to 5 years.

Before your blood and tumor samples can be used for research, the people doing the research must get specific approval from the institutional review board (IRB) of M. D. Anderson. The IRB is a committee made up of doctors, researchers, and members of the community. The IRB is responsible for protecting the participants involved in research studies and making sure all research is done in a safe and ethical manner. All research done at M. D. Anderson, including research involving your blood and/or tumor samples from this bank, must first be approved by the IRB.

This is an investigational study. Up to 200 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a suspected or confirmed diagnosis of malignant melanoma. These include patients with melanoma of the soft part, spindle-cell neoplasm consistent with melanoma and choroidal melanoma.
2. Patients who are willing to consent for this protocol.

Exclusion Criteria: None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants with a diagnosis of malignant melanoma.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2006-06-13 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Collection and long-term collection of blood and tumor samples from patients with malignant melanoma for future biological and/or surrogate marker studies. | 6 Years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Davies, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org